CLINICAL TRIAL: NCT00545428
Title: Mastoid Bone Autograft for Dorsal Nasal Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Lucas Gomes Patrocinio, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Patrocinio
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Nose Deformities, Acquired
Keywords: Nasal acquired diseases; Nasal congenital diseases; Rhinoplasty; Grafts
MeSH Terms: conditions — Nose Deformities, Acquired | interventions — Rhinoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Rhinoplasty
  Interventions: Procedure: Rhinoplasty

INTERVENTIONS:
Procedure: Rhinoplasty — Mastoid bone autograft for dorsal nasal augmentation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mastoid bone autograft for dorsal nasal augmentation in rhinoplasty.

DETAILED DESCRIPTION:
INTRODUCTION: Several grafts and/or implants have been used for dorsal augmentation. In some cases, especially the traumatic, non-caucasian, and multi-operated ones, the amount of augmentation is higher than the usually available from septal and auricular conchal autografts.

OBJECTIVE: To evaluate the safety and efficacy of mastoid bone autograft for dorsal nasal augmentation in rhinoplasty.

DESIGN: A prospective study of 15 consecutive patients submitted to dorsal nasal augmentation with mastoid bone, during a 2-year period.

SETTING: One major academic medical center.

ELIGIBILITY:
Inclusion Criteria:

* Nasal acquired or congenital deformity of the dorsum that requires augmentation of more than 5 mm

Exclusion Criteria:

* Previous otologic surgery/disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction | 1 year

SECONDARY OUTCOMES:
Observer's satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lucas G Patrocinio, MD, Principal Investigator — Federal University of Uberlandia, Department of ENT/H&N; Jose A Patrocinio, MD, PhD, Study Chair — Federal University of Uberlandia, Department of ENT/H&N
Locations (1):
- Federal University of Uberlandia, Department of ENT/H&N, Uberlândia, Minas Gerais, Brazil

REFERENCES:
- [Background] Baser B, Shahani R, Khanna S, Grewal DS. Calvarial bone grafts for augmentation rhinoplasty. J Laryngol Otol. 1991 Dec;105(12):1018-20. doi: 10.1017/s0022215100118109. PMID 1787353
- [Background] Jovanovic S, Berghaus A. Autogenous auricular concha cartilage transplant in corrective rhinoplasty. Practical hints and critical remarks. Rhinology. 1991 Dec;29(4):273-9. PMID 1780628
- [Background] Patrocinio LG, Patrocinio JA. Open rhinoplasty for African-American noses. Br J Oral Maxillofac Surg. 2007 Oct;45(7):561-6. doi: 10.1016/j.bjoms.2007.01.011. Epub 2007 Mar 12. PMID 17350737
- [Background] Pedroza F, Anjos GC, Patrocinio LG, Barreto JM, Cortes J, Quessep SH. Seagull wing graft: a technique for the replacement of lower lateral cartilages. Arch Facial Plast Surg. 2006 Nov-Dec;8(6):396-403. doi: 10.1001/archfaci.8.6.396. PMID 17116787
- [Background] Patrocinio LG, Carvalho PM, de Souza HM, Couto HG, Patrocinio JA. Surgical maneuvers performed on rhinoplasty procedures carried out at an otorhinolaryngology residency program. Braz J Otorhinolaryngol. 2006 Jul-Aug;72(4):439-42. doi: 10.1016/s1808-8694(15)30986-1. PMID 17143420